CLINICAL TRIAL: NCT05019391
Title: Clinical and Radiological Evaluation of Patients With Vertebrobasilar Insufficiency in Assiut University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMohamed, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: vertebrobasilar insufficiency
Record Dates: First submitted 2021-08-16; First posted 2021-08-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Vertebrobasilar Insufficiency
Keywords: vertebrobasilar-insufficiency-transcranial-doppler
MeSH Terms: conditions — Vertebrobasilar Insufficiency | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: A cohort study will be performed on at least 100 patients presented with vertebrobasilar insufficiency including vertebrobasilar stroke or vertebrobasilar TIA who will be admitted in department of neurology in assiut university hospital.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transcranial doppler — it provides an accurate, noninvasive, and simple method for the diagnosis of VBI. Through the diagnosis results, it will be clear about the blood flow status of single vessel and vascular compliance, which is helpful for accurate reflection of the subtle changes of VBI

SUMMARY:
Clinical and radiological evaluation including transcranial Doppler of vertebral arteries of patients with vertebrobasilar insufficiency attending assiut university hospital and assessment of possible risk factors that may lead to vertebrobasilar insufficiency.

DETAILED DESCRIPTION:
Vertebrobasilar insufficiency (VBI) is defined by inadequate blood flow through the posterior circulation of the brain, supplied by the 2 vertebral arteries that merge to form the basilar artery. Transient ischemic attacks in the vertebrobasilar system represent 20% of all transient ischemic attacks, Their diagnosis is more difficult than that of ischemic attacks in the anterior circulation because its manifestations are subjective and difficult to quantify. Although traditionally VB stroke is regarded as having a more benign outcome when compared to anterior circulation stroke, data is still conflicting, with some studies showing a higher impairment in VB stroke patients with 21% of death or major disability at 3 months. Transient ischemic attacks and, more rarely, infarcts in the posterior circulation may be due to subclavian steal syndrome. Basilar artery transient ischemic attacks usually occur after the six decade, syncopal attacks occur in about 10% sudden in onset and brief in duration. Regarding the clinical presentation of VB stroke, the common symptoms are dizziness, unilateral limb weakness, headache, vomiting and nausea; as for clinical signs, the most frequent are unilateral limb weakness, gait ataxia, unilateral limb ataxia, dysarthria and nystagmus. Previously, there was no simple and effective method for the detection of VBI, but in recent years, with the development and progress of medical technology and the emergence of Transcranial Doppler (TCD), it provides an accurate, noninvasive, and simple method for the diagnosis of VBI. Through the diagnosis results, it will be clear about the blood flow status of single vessel and vascular compliance, which is helpful for accurate reflection of the subtle changes of VBI.

ELIGIBILITY:
Inclusion Criteria:

1. patients with vertigo of central origin, syncopal attacks, frequent imbalance that not related to aural origin.
2. clinical examination and imaging (MRI or CT) with the diagnosis standard of vertebrobasilar insufficiency including vertebrobasilar stroke and vertebrobasilar TIA.
3. patients with abnormal lipogram and cervical spondylosis
4. patients aged > 45 years old of both sex.

Exclusion Criteria:

1. subjective complain of aural vertigo or test to exclude aural vertigo.
2. patients with malignant tumor.
3. pregnant or lactating women.
4. cognitive impairment and mental illness.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Detection and estimation of risk factors for vertebrobasilar insufficiency patients | 3 years
  Evaluation and detection of possible risk factors that may lead to vertebrobasilar insufficiency by using Doppler ultrasound and detection of rate of vertebrobasilar insufficiency due to central vertigo or frequent imbalance attacks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caplan L, Chung CS, Wityk R, Glass T, Tapia J, Pazdera L, Chang HM, Dashe J, Chaves C, Vemmos K, Leary M, Dewitt L, Pessin M. New England medical center posterior circulation stroke registry: I. Methods, data base, distribution of brain lesions, stroke mechanisms, and outcomes. J Clin Neurol. 2005 Apr;1(1):14-30. doi: 10.3988/jcn.2005.1.1.14. Epub 2005 Apr 30. PMID 20396469